CLINICAL TRIAL: NCT00382850
Title: Randomized Controlled Trial of Laparoscopic Compared to Open Nissen Fundoplication in Children Younger Than 2 Years of Age
Brief Title: Clinical Trial Comparing Open and Laparoscopic Nissen Fundoplication in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-08-01-01
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Gastroesophageal Reflux
Keywords: Nissen fundoplication; gastroesophageal reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Fundoplication

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- open nissen fundoplication (Active Comparator): open repair through surgical midline incision
  Interventions: Procedure: Nissen fundoplication
- laparoscopic nissen fundoplication (Active Comparator): use of laparoscope to do repair
  Interventions: Procedure: Nissen fundoplication

INTERVENTIONS:
Procedure: Nissen fundoplication

SUMMARY:
The purpose of this study is to determine whether short- and long-term outcomes are different between open and laparoscopic Nissen fundoplication performed in children younger than 2 years of age.

DETAILED DESCRIPTION:
Nissen fundoplication is a commonly performed procedure in infants and children with gastroesophageal reflux and a variety of other medical conditions including respiratory compromise, severe neurologic impairment, failure to thrive and swallowing dysfunction. Randomized controlled trials in adults have shown that laparoscopic fundoplication is a safe procedure that results in lower morbidity, shorter hospital length of stay and similar 5-year recurrence rates when compared to an open procedure. The aim of this study is to compare laparoscopic and open Nissen fundoplication in children less than 2 years of age.

Children younger than 2 years of age presenting for Nissen fundoplication will be randomized to either a laparoscopic or an open procedure. Patients who have already undergone anti-reflux surgery or whose hospitalization is anticipated to be prolonged by an unrelated illness will be excluded. All procedures will be performed at a single institution by two surgeons who will perform both the open and laparoscopic procedures.

A total of 68 patients will be needed (34 in each group) to detect a 20% difference in length of stay at a significance level of p < 0.05 and power of 80%. Patients will be followed for up to 2 years postoperatively. Variables to be compared between the two groups will include age, gender, presence of neurologic impairment, presence and specification of any congenital abnormalities, total operative time, total dose of narcotic analgesia required, postoperative day on which the patient tolerated full feedings, postoperative and total lengths of stay as well as the occurrence of postoperative complications (including wound infection and the need for immediate reoperation). The primary outcomes analyzed will be length of stay and amount of narcotic analgesia required. Longer-term outcomes including persistent GERD, wrap failure and need for reoperation within 24 months of the initial procedure also will be determined.

ELIGIBILITY:
Inclusion Criteria:

* clinical or radiographic diagnosis of gastroesophageal reflux
* age less than 2 years (24 months) at the time of surgery

Exclusion Criteria:

* prior fundoplication procedure
* concomitant need for an intraabdominal procedure (except gastrostomy tube placement)
* esophageal dysmotility
* hospitalization expected to be prolonged due to a concurrent illness actively being treated (e.g. congenital heart disease requiring surgical repair during the same hospitalization)

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2005-11; Primary Completion 2010-11-30 (Actual); Study Completion 2010-11-30 (Actual)

PRIMARY OUTCOMES:
postoperative length of stay | 0 to 14days
  days in hospital
postoperative narcotic pain medication requirements | 0 to 14 days
  days requiring narcotics for pain relief
length of time to tolerating full feeds prior to discharge | 0 to 7 days
  days after surgery before feeding begins

SECONDARY OUTCOMES:
intraoperative complication rates | duration of procedure
  complications of procedure
wrap failure and need for subsequent reoperation | up to 2 yrs
  operative failure
need for continued medical therapy for GER | up to 2 yrs
  symptomatic reflux requiring medication
death | up to 2 years
  death

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Colombani, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States